CLINICAL TRIAL: NCT01256606
Title: Investigational Study of a Prenatal Diagnostic Test for Fetal Aneuploidy
Brief Title: Prenatal Test for Fetal Aneuploidy Detection
Status: Completed | Type: Observational
Sponsor: Roche Sequencing Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: TT001
Record Dates: First submitted 2010-11-22; First posted 2010-12-08 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Aneuploidy; Trisomy 21
MeSH Terms: conditions — Aneuploidy; Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive for fetal aneuploidy
- Negative for fetal aneuploidy

SUMMARY:
The purpose of this study is to develop and evaluate a blood test for pregnant women for detection of fetal aneuploidy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18yrs or older
* Subject has a singleton pregnancy
* Subject is planning to undergo chorionic villus sampling (CVS) and/or amniocentesis with current pregnancy
* Subject is able to provide consent

Exclusion Criteria:

* Subject is pregnant with more than one fetus
* Subject (mother) has known aneuploidy
* Subject has active malignancy requiring major surgery or systemic chemotherapy or has a history of metastatic cancer.
* Subject has already undergone CVS or amniocentesis during current pregnancy prior to study enrollment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women planning to undergo chorionic villus sampling or amniocentesis for fetal genetic evaluation
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2010-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Comparison of blood test to results from chorionic villus sampling or amniocentesis for fetal aneuploidy detection | 24 months
  Circulating genomic material from maternal blood will be quantified using biochemical techniques to determine the presence of fetal aneuploidy. The results obtained from analysis of circulating genomic material will be compared to the karyotype results from chorionic villus sampling or amniocentesis.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Song, MD, Study Director — Ariosa Diagnostics
Locations (6):
- United States (6):
  - East Bay Perinatal Medical Associates, Oakland, California
  - Prenatal Diagnosis of Northern California, Sacramento, California
  - University of California - San Diego, San Diego, California
  - University of California - San Francisco, San Francisco, California
  - Atlanta Perinatal Consultants, Atlanta, Georgia
  - Medical College of Wisconsin, Milwaukee, Wisconsin